CLINICAL TRIAL: NCT00950638
Title: A Phase I Study to Establish the Safety and Tolerability of ARC1905 (Anti-C5 Aptamer) in Subjects With Dry Age-related Macular Degeneration
Brief Title: A Study of ARC1905 (Anti-C5 Aptamer) in Subjects With Dry Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPH2001
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Dry Age-Related Macular Degeneration
Keywords: AMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dose comparison (Active Comparator)
  Interventions: Drug: Avacincaptad Pegol
- Dose comparison (Active Comparator)
  Interventions: Drug: Avacincaptad Pegol

INTERVENTIONS:
Drug: Avacincaptad Pegol — intravitreal injection
  Other Names: Zimura (previous name); IZERVAY; ARC1905

SUMMARY:
The objectives of this study are to evaluate the safety and tolerability of ARC1905 intravitreous injection in subjects with geographic atrophy secondary to dry age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

Dry AMD (drusen and/or geographic atrophy) in both eyes

Exclusion Criteria:

* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication.

Any ocular or periocular infection (including blepharitis), or ocular surface inflammation in the past twelve (12) weeks.

History of any of the following procedures: Posterior vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant or retinal detachment.

Any of the following underlying diseases including:

* Diabetic retinopathy
* History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV ), history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within last 6 months, ventricular tachyarrythmias requiring ongoing treatment.
* History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.
* Clinically significant impaired renal (serum creatinine >2.5 mg/dl or status post renal transplant or receiving dialysis) or hepatic function. Subjects with results outside these ranges may be enrolled in consultation with Ophthotech.
* Stroke (within 12 months of trial entry).
* Any major surgical procedure within one month of trial entry. Previous therapeutic radiation in the region of the study eye. Any treatment with an investigational agent in the past 60 days for any condition.

Women who are pregnant or nursing. Known serious allergies to the fluorescein dye used in angiography or to the components of the ARC1905 formulation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-07-16 (Actual); Primary Completion 2011-03-24 (Actual); Study Completion 2011-03-24 (Actual)

PRIMARY OUTCOMES:
Presence of any dose-limiting toxicity (DLT), safety endpoints include adverse events, vital signs, ophthalmic variables and outcomes | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthotech, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26394&tenant=MT_AST_9011